CLINICAL TRIAL: NCT06326983
Title: Opioid Sparing Anesthesia Care for Pediatric Patients Having Tonsil Surgery; a Randomized, Controlled, Non-inferiority Study
Brief Title: Opioid Sparing Anesthesia Care for Pediatric Patients Having Tonsil Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Arielle Mizrahi-Arnaud, MD, Anesthesia, Critical Care and Pain Medicine, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00047028
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Tonsillitis; Post-operative Nausea and Vomiting (PONV); Emergence Delirium; Opioid Analgesic Adverse Reaction; Anesthesia; Pain
MeSH Terms: conditions — Tonsillitis; Vomiting; Emergence Delirium; Pain | interventions — Dexmedetomidine; Acetaminophen; Ketorolac; Ketorolac Tromethamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-Sparing Anesthetic Plan (Experimental): For their tonsil surgery, subjects will receive Dexmedetomidine (1mcg/kg bolus given intravenously at induction of anesthesia) and Acetaminophen (12.5mg/kg with a maximum dose of 1 gram given intravenously at induction of anesthesia). Ketorolac 0.5mg/kg with a max dose of 30mg given intravenously at the end of surgery. No opioids will be given during the procedure.
  Interventions: Drug: Dexmedetomidine; Drug: Acetaminophen; Drug: Ketorolac
- Opioid Anesthetic Plan (Active Comparator): For their tonsil surgery, subjects will receive Morphine (0.1mg/kg given intravenously at induction of anesthesia) and Acetaminophen (12.5mg/kg with a maximum dose of 1 gram given intravenously at induction of anesthesia). Ketorolac 0.5mg/kg with a max dose of 30mg intravenously at the end of surgery.
  Interventions: Drug: Acetaminophen; Drug: Ketorolac; Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (1mcg/kg bolus given intravenously at induction of anesthesia
  Other Names: Precedex
  Arms: Opioid-Sparing Anesthetic Plan
Drug: Acetaminophen — Acetaminophen (12.5mg/kg with a maximum dose of 1 gram given intravenously at induction of anesthesia).
  Other Names: Ofirmev
Drug: Ketorolac — Ketorolac 0.5mg/kg with a max dose of 30mg intravenously at the end of surgery.
  Other Names: Toradol
Drug: Morphine — Morphine (0.1mg/kg given intravenously at induction of anesthesia)
  Arms: Opioid Anesthetic Plan

SUMMARY:
This is a prospective, randomized, controlled, non-inferiority study of patients undergoing tonsil surgeries at Boston Children's Hospital Waltham. The overall aim is to evaluate the efficacy of an opioid anesthetic plan (morphine, ketorolac, and acetaminophen versus an opioid sparing anesthetic plan (dexmedetomidine, ketorolac and acetaminophen) for perioperative analgesia and recovery time in patients undergoing tonsillectomies and tonsillotomies at Boston Children's Hospital Waltham. Secondary measures include rescue opioids administered in post-anesthesia care unit (PACU), re-operation secondary to bleeding, emergence delirium, post-operative nausea and vomiting, intraoperative hemodynamics, intraoperative vasopressor administration, and length of procedure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia classification status I-III
* Ages 3 years to 17 years
* Scheduled for tonsillectomy or tonsillotomy with or without adenoidectomy at Boston Children's Hospital Waltham

Exclusion Criteria:

* Patients not scheduled for primary tonsillectomy/tonsillotomy.
* Patients with known coagulopathies
* Patients with previous chronic pain syndromes
* Patients with any condition/indication that would prevent them from being able to be randomized (i.e. allergy to one of the study medications)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Median Pain Scores in the Post-Anesthesia Care Unit | entry to post-anesthesia care unit to 2-6 hours post-operatively
  Median Pain Scores in the Post-Anesthesia Care Unit measured by the numeric rating scale (NRS), Wong-Baker Faces scale or FLACC (Face, Legs, Activity, Cry, Consolability) scale as indicated based on patient age and development. All scales are done on a 0-10 point scale with 0 being no pain and 10 being the highest pain.
Post-operative pain at 12-24 hours | 12-24 hours post-operatively
  Pain categorized as none, mild, moderate, and severe. Taken from the routine follow-up nursing phone call.
Post Operative Anesthesia Unit Length of Stay (hours) | From entry to the Post Anesthesia Care Unit to exit from the Post-Anesthesia Care Unit. Assessed for up to 8 hours on the date of surgery
  Length of time spent in the Post Operative Anesthesia Unit after tonsil surgery

SECONDARY OUTCOMES:
Opioid rescue medication administration | surgery end to 2-6 hours post-operatively
  Opioid rescue medications administered (reported as oral morphine equivalents)
Emergence Delirium | surgery end to 2-6 hours post-operatively
  Incidence of emergence delirium defined as a score ≥ 10 on the Pediatric Anesthesia Emergence Delirium Scale. Scores range 0-20 with 0 being no agitation/delirium to 20 being the highest level.
Post-operative nausea and vomiting | surgery end to 2-6 hours post-operatively
  Incidence of episodes of emesis or administration of anti-emetics in the post-anesthesia care unit
Procedure length (minutes) | 0-60 minutes
  from incision time to patient being wheeled out of the operating room
Intraoperative Blood pressure (mmHg) | 10 minutes
  Range of systolic blood pressure within 10 minutes of anesthesia induction
Intraoperative Heart rate (beats per second) | 10 minutes
  Range of heart rate within 10 minutes of anesthesia induction
Vasopressor administration | 0-60 minutes
  Intraoperative administration of vasopressors

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No